CLINICAL TRIAL: NCT00374192
Title: The Treatment of Insomnia in Symptomatic Peri- and Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Lee S. Cohen, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-P000194
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-08

CONDITIONS: Menopause; Insomnia
Keywords: Menopause; Insomnia; Depression; Anxiety; Sleep; Lunesta; Quality of Life
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Anxiety Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Eszopiclone
  Interventions: Drug: Eszopiclone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone — 3 mg per day
  Other Names: Lunesta
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
To examine the change in sleep patterns and mood symptoms in response to eszopiclone (Lunesta) using a double-blind placebo-controlled cross-over study design in perimenopausal and postmenopausal women who experience insomnia, mild depression and/or anxiety.

DETAILED DESCRIPTION:
The study design is a double-blinded placebo-controlled cross-over study that will be completed at the MGH site. It is an 11-week study of insomnia, mild mood, and anxiety symptoms in peri- and postmenopausal women age 40 years or older. Subjects who are enrolled will have 5 office visits during the 11-week long study.

Various studies have identified female gender as a strong risk factor for insomnia, (Ford & Kamerow, 1989; Klink et al, 1992; Li et al, 2002);community-based studies that examined gender differences in insomnia complaints have consistently shown a higher prevalence of insomnia among women than among men. It has been hypothesized that insomnia might be an overlooked complaint among women seeking treatment in the primary care setting.

Insomnia and other sleep disturbances may be reported during specific situations associated with the female reproductive cycle, such as pregnancy (Sahota et al, 2003) and menopause (Joffe et al, 2003). Complaints of sleep-onset and sleep-maintenance insomnia are among the most common symptoms in peri- and postmenopausal women. This sleep disturbance frequently co-occurs with hot flushes and depression symptoms. The menopausal transition is also a period of heightened vulnerability to mood and anxiety disturbances, and significant vasomotor symptoms (i.e. hot flushes and night sweats) which may affect functioning and quality of life.

Consented subjects will track their sleep patterns for one week using a sleep diary to confirm that they have either difficulty initiating sleep (³ 30 minutes) or difficulty maintaining sleep (wake time after sleep onset ³ 30), for ≥ 3 nights during 7-day observation period. Those who are confirmed to meet these insomnia criteria will be randomized in a 1-to-1 fashion to cross-over treatment starting with either eszopiclone or placebo.

In addition to taking the daily medication, and coming to the office visits, subjects will complete a daily diary throughout the study. This diary is completed to assess insomnia symptoms throughout the duration of the study. Treatment assignments will be revealed at final study visit to the participant, research coordinator, and study physician.

ELIGIBILITY:
Inclusion Criteria:

1. Women 40+ years old.
2. Subject must have any of the following perimenopausal or postmenopausal signs and symptoms as defined by the Stages of Reproductive Aging Workshop (STRAW):

   1. Early Menopausal Transition (Stage -2): Variable cycle length >7 days different from normal.
   2. Late Menopausal Transition (Stage -1) : > 2 skipped cycles and an interval of amenorrhea > 60 days.
   3. Post Menopause (Stage +1): Amenorrhea for at least 12 months.
   4. Surgical Post Menopause
   5. Hysterectomized women with one or both ovaries preserved will be eligible if FSH levels > 20 IU/L.
   6. If on hormonal therapy, history of menstrual-cycle abnormalities consistent with any of 2a-2e above indicating peri-/postmenopausal status prior to initiation of hormonal therapy.
3. One or both the following insomnia symptoms for ³ 3 nights per week for at least one month prior to study enrollment:

   1. Difficulty initiating sleep (³ 30 minutes)
   2. Difficulty maintaining sleep (wake time after sleep onset ³ 30 minutes)
4. Daytime function or well-being is impaired as a result of insomnia.
5. Mild depression and/or anxiety at screening visit defined as:

   1. Mild Depressive symptoms defined by Montgomery-Åsberg Depression Rating Scale-MADRS (MADRS) ³ 10 administered at screening visit, or
   2. Mild Anxiety symptoms defined by Beck Anxiety Inventory (BAI) ³ 10 administered at screening visit.
6. May have (but not required) hot flushes
7. May have (but not required) developed insomnia after discontinuation of hormonal therapy.
8. If subject is on an antidepressant, they must have stable doses for at least 2 months.
9. If subject is on hormonal therapy, dose must be stable for at least 2 months.
10. General Good Health

Exclusion Criteria:

1. According to M.I.N.I (Mini International Neuropsychiatric Interview), subject meets current or past criteria for past 3 months:

   1. Major Depression
   2. Dysthymia
   3. Panic disorder
   4. PTSD (Post-Traumatic Stress Disorder)
2. According to M.I.N.I, subject has no evidence of current suicidal ideation, homicidal ideation, or psychotic symptoms at screening visit.
3. Suicide attempt in the past 5 years.
4. According to M.I.N.I, subject meets criteria for substance use disorder diagnosis within the past 5 years.
5. Subject has current or recent use (in the past month and used > 25% of time) of hypnotic agents.
6. Subject is on an antidepressant or hormone therapy in past 2 months. (Unless they are taking currently and have had a stable dose for ≥ 2 months).
7. Subject has:

   1. Unstable medical abnormality
   2. Unstable chronic disease.
8. History of significant cardiac, renal, or hepatic disease, or seizure disorder.
9. Regular use of any disallowed medication (Including; Clarithromycin, Itraconazole, Ketoconazole, Nefazodone, Nelfinavir, Olanzapine, Rifampin, Ritonavir, Troleandomycin) currently or in the past month.
10. Subject has a disorder or history of a condition (e.g., mal-absorption, gastrointestinal surgery) that may interfere with drug absorption, distribution, metabolism, or excretion.
11. Subject has a been previously diagnosed sleep apnea, restless leg syndrome (RLS), or periodic leg movement syndrome (PLMS), or has any condition that may affect sleep (e.g., chronic pain, urinary incontinence, etc.).
12. Subject reports consumption of more than two alcoholic beverages daily, 14 or more alcoholic beverages weekly, or five or more alcoholic beverages on any given day during the past month.
13. Currently pregnant or breastfeeding
14. Subject is a rotating or third/night shift worker.
15. Subject often travels across multiple time zones.
16. Subject is currently enrolled in another clinical trial, subject has participated in any investigational drug study within 30 days prior to screening, or plans to participate in another investigational drug study during participation in this study.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To examine the effect of treatment with eszopiclone on sleep-onset and sleep-maintenance insomnia in peri- and postmenopausal women. | 4 weeks

SECONDARY OUTCOMES:
To examine the effect of eszopiclone on mood and quality of life in peri- and postmenopausal women with insomnia who have comorbid depressive and/or anxiety symptoms. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lee S. Cohen, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: MGH Center for Women's Mental Health — http://www.womensmentalhealth.org